CLINICAL TRIAL: NCT05372653
Title: A Phase 3, Multicenter, Open-label, Uncontrolled Trial to Evaluate the Efficacy and Safety of OPA-15406 Ointment in Infants Younger Than 2 Years of Age With Atopic Dermatitis
Brief Title: A Long-term Trial of OPA-15406 in Infants With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 271-102-00016
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPA-15406 (Experimental)
  Interventions: Drug: OPA-15406

INTERVENTIONS:
Drug: OPA-15406 — 0.3% or 1% ointment, topical, twice daily, for 52 weeks
  Other Names: difamilast

SUMMARY:
To investigate the efficacy of 0.3% OPA-15406 ointment when administered twice daily for 4 weeks in infants younger than 2 years of age with Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are diagnosed with AD in accordance with the criteria of the Japanese Dermatological Association
* Subjects whose AD affects 5% to 40% of BSA (excluding scalp) at the screening and baseline examinations
* Subjects who have an IGA score of 2 or 3 at the screening and baseline examinations

Exclusion Criteria:

-Subjects who have an AD or contact dermatitis flare-up defined as a rapid intensification of AD, within 28 days prior to the baseline examination

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Sotobo Children's Clinic, Isumi, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

REFERENCES:
- [Derived] Saeki H, Ohya Y, Baba N, Imamura T, Yokota D, Tsubouchi H. A Phase 3, Long-Term, Open-Label Study of Difamilast Ointment to Evaluate Efficacy and Safety in Japanese Infants with Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Oct 31. doi: 10.1007/s13555-025-01581-1. Online ahead of print. PMID 41171590
- [Derived] Saeki H, Ohya Y, Baba N, Imamura T, Yokota D, Tsubouchi H. An Interim Report of a Phase 3, Long-Term, Open-Label Study to Evaluate Efficacy and Safety of Difamilast Ointment in Japanese Infants with Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2443-2455. doi: 10.1007/s13555-024-01236-7. Epub 2024 Jul 29. PMID 39075274

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3% OPA-15406: The 0.3% formulation was topically administered twice daily (approximately 12 hours apart between morning and night administrations) for 52 weeks.
- 1% OPA-15406: As the starting dose, the 0.3% formulation was topically administered twice daily (approximately 12 hours apart between morning and night administrations) . After 4 weeks of the IMP administration, the 1% formulation was administered twice daily in accordance with the prespecified rules for dose increase.
Period: Overall Study
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Started | 12 | 29
Completed | 11 | 25
Not Completed | 1 | 4
Not completed — Study treatment terminated by parent/guardian | 1 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Total
Number analyzed (Participants) | 12 | 29 | 41
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.9 (3.9) | 10.8 (5.4) | 10.0 (5.1)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: <12 months | 10 | 18 | 28
  Age Group: >=12 months | 2 | 11 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 7 | 19 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 12 | 29 | 41
Region of Enrollment [Number; unit: participants]
  Japan | 12 | 29 | 41

OUTCOME MEASURES:

1. Primary Outcome: Success Rate in IGA (Percentage of Subjects With an IGA Score of 0 or 1 With Improvement by at Least 2 Grades)
Description: The investigator or sub investigator assessed the skin symptoms using IGA (Investigator's Global Assessment). The investigator or sub investigator scored the severity (0 = clear, 1 = almost clear, 2 =mild, 3 = moderate, 4 = severe/very severe) of the overall symptoms of the treatment area (erythema, infiltration, papules, effusion and scab formation) from baseline to Week 4. Incidence of success in IGA was defined as the rate of subjects whose IGA score is 0 (clear) or 1 (almost clear) and had improved by at least 2 grades (responders) from baseline.
Time Frame: Week 4
Population: The efficacy analysis set (FAS [full analysis set]) consisted of all subjects who received the IMP at least once.
Measure: Number (95% Confidence Interval); unit: Percentage of perticipants
Arm/Group | 0.3% OPA-15406
Number analyzed (Participants) | 41
Percentage of perticipants | 56.10 [39.75 to 71.53]

2. Secondary Outcome: Response Rate in Eczema Area and Severity Index (EASI) 75 (Improvement of ≥75% in EASI)
Description: Response (improvement) in EASI 75 was defined as a decrease by ≥75% in the percent change from baseline in the total score of EASI.
Time Frame: Week4
Population: The efficacy analysis set (FAS [full analysis set]) consisted of all subjects who received the IMP at least once.
Measure: Number (95% Confidence Interval); unit: Percentage of perticipants
Arm/Group | 0.3% OPA-15406
Number analyzed (Participants) | 41
Percentage of perticipants | 82.93 [67.94 to 92.85]

ADVERSE EVENTS:
Time Frame: Adverse event collection begins after a legal guardian signs the ICF, and continues until the completion of the 52-week follow-up examination (or the final observation day).
Description: The safety analysis set (SS) consisted of all subjects who received the IMP at least once.
  The groups were described separately to identify adverse events that occurred in the subjects who had received only the 0.3% formulation and those that occurred in the subjects who had received the 1% formulation at least once.
Groups:
- 0.3% OPA-15406: The 0.3% formulation was topically administered twice daily (approximately 12 hours apart between morning and night administrations) .
  In this section, we display the adverse events that occurred at the time of administration of the 0.3% formulation.
- 1% OPA-15406: After 4 weeks of the 0.3% formulation administration, the 1% formulation was administered twice daily in accordance with the prespecified rules for dose increase.
  In this section, we display the adverse events that occurred at the time of administration of the 1.0% formulation.
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/29
Other Adverse Events (participants affected / at risk) | 24/41 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% OPA-15406 (N=41) | 1% OPA-15406 (N=29)
Kawasaki's disease (Vascular disorders) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% OPA-15406 (N=41) | 1% OPA-15406 (N=29)
Conjunctivitis allergic (Eye disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 3
Bronchitis (Infections and infestations) | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 2
Croup infectious (Infections and infestations) | 0 | 2
Folliculitis (Infections and infestations) | 0 | 5
Gastroenteritis (Infections and infestations) | 4 | 16
Gastroenteritis viral (Infections and infestations) | 0 | 2
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 5
Herpangina (Infections and infestations) | 0 | 4
Impetigo (Infections and infestations) | 3 | 3
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 18 | 24
Otitis media (Infections and infestations) | 0 | 2
Otitis media acute (Infections and infestations) | 0 | 8
Pharyngitis (Infections and infestations) | 0 | 4
Rhinitis (Infections and infestations) | 0 | 2
Skin candida (Infections and infestations) | 0 | 3
Adenovirus infection (Infections and infestations) | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 3 | 2
Conjunctivitis bacterial (Infections and infestations) | 0 | 6
Metapneumovirus infection (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 4 | 7
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 4
Scratch (Injury, poisoning and procedural complications) | 0 | 2
Mouth injury (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Lip injury (Injury, poisoning and procedural complications) | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Balanoposthitis (Reproductive system and breast disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 8 | 8
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 10
Miliaria (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT05372653/Prot_SAP_000.pdf